CLINICAL TRIAL: NCT01534884
Title: Phase 1, Randomized, Controlled, Multicenter, 2-Arm, Parallel-Group, Double-Blind Study to Demonstrate the Equivalence of CT-P10 to MabThera With Respect to the Pharmacokinetic Profile in Patients With Rheumatoid Arthritis
Brief Title: Demonstrate the Equivalence of CT-P10 to MabThera With Respect to the Pharmacokinetic Profile in Patients With Rheumatoid Arthritis
Acronym: Triad RA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-P10 1.1; 2011-002822-37 (EudraCT Number)
Record Dates: First submitted 2012-02-08; First posted 2012-02-17 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
Keywords: RA, Biosimilar
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MabThera (Active Comparator): rituximab
  Interventions: Biological: rituximab
- CT-P10 (Active Comparator): rituximab
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab — 1000 mg by intravenous (IV) infusion. Each patient may receive 2 courses of treatment.

SUMMARY:
This randomized,controlled, multicenter, 2-arm, parallel-group, double-blind, prospective, Phase 1 study is designed to demonstrate comparable pharmacokinetics in terms of AUC0-last and Cmax (after second infusion) between CT-P10 and MabThera in patients with active RA concomitantly treated with MTX during the Core Study Period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a diagnosis of RA according to the revised 1987 ACR classification criteria (Arnett et al 1987) for at least 6 months prior to randomization.
2. Patient has active disease as defined by the presence of 6 or more swollen joints (of 66 assessed) and 6 or more tender joints (of 68 assessed), and serum CRP ≥1.5 mg/dL or an ESR ≥28 mm/hour.

Exclusion Criteria:

1. Patient is unresponsive or intolerable to more than 2 biologic agents.
2. Patient has allergies or hypersensitivity to murine, chimeric, human, or humanized proteins.
3. Patient has current or past history of chronic infection with hepatitis B, hepatitis C, or infection with human immunodeficiency virus (HIV)-1 or -2 or who has a positive result to the screening test for these infections.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
PK in terms of Cmax | Up to Week 24
  maximum serum concentration

CONTACTS AND LOCATIONS:
Overall Officials: DaeHyun Yoo, M.D., Ph.D., Study Director — Hanyang University
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Yoo DH, Suh CH, Shim SC, Jeka S, Molina FFC, Hrycaj P, Wiland P, Lee EY, Medina-Rodriguez FG, Shesternya P, Radominski S, Stanislav M, Kovalenko V, Sheen DH, Myasoutova L, Lim MJ, Choe JY, Lee SJ, Lee SY, Kim SH, Park W. Efficacy, Safety and Pharmacokinetics of Up to Two Courses of the Rituximab Biosimilar CT-P10 Versus Innovator Rituximab in Patients with Rheumatoid Arthritis: Results up to Week 72 of a Phase I Randomized Controlled Trial. BioDrugs. 2017 Aug;31(4):357-367. doi: 10.1007/s40259-017-0232-7. PMID 28612179
- [Derived] Yoo DH, Suh CH, Shim SC, Jeka S, Cons-Molina FF, Hrycaj P, Wiland P, Lee EY, Medina-Rodriguez FG, Shesternya P, Radominski S, Stanislav M, Kovalenko V, Sheen DH, Myasoutova L, Lim MJ, Choe JY, Lee SJ, Lee SY, Kwon TS, Park W. A multicentre randomised controlled trial to compare the pharmacokinetics, efficacy and safety of CT-P10 and innovator rituximab in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Mar;76(3):566-570. doi: 10.1136/annrheumdis-2016-209540. Epub 2016 Sep 13. PMID 27624791